CLINICAL TRIAL: NCT00238524
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of 400mg/Day and 600mg/Day SPM 927 (Lacosamide) in Subjects With Painful Distal Diabetic Neuropathy
Brief Title: A Trial to Assess the Efficacy and Safety of SPM 927 (Lacosamide) in Subjects With Painful Distal Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0743
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2010-04

CONDITIONS: Diabetic Neuropathy
Keywords: painful distal diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

INTERVENTIONS:
Drug: SPM 927

SUMMARY:
This trial was conducted at about 50 sites in Europe and has been clinically completed. Patients had symptoms of painful diabetic neuropathy for 6 months up to 5 years with an optimized diabetic control and at least moderate pain. Patients were not eligible with other chronic pain or any other medical or psychiatric condition, that would have jeopardized or compromised the patient's ability to participate in the trial. After a 2-week run-in phase patients were randomly assigned to one of three treatment arms. All patients who had completed the 6-week titration phase to reach their target dose entered a 12-week maintenance phase. At the end of the maintenance phase, subjects were offered the option of entering the open-label, follow-on trial. The change in pain was measured daily as well as interference of pain with sleep and general activity.

ELIGIBILITY:
Inclusion Criteria:

* Painful distal diabetic neuropathy

Exclusion Criteria:

* Symptoms of painful distal diabetic neuropathy for less than six months or greater than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2003-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Investigate the efficacy of lacosamide compared with placebo in reducing pain in subjects with painful distal diabetic neuropathy will be determined by pain score ratings assessed in a patient's diary and at clinic visits.

SECONDARY OUTCOMES:
Investigate effect of lacosmide on subjects' perception of sleep, activity, quality of life, and safety, determined by rating scales assessed in a patient's diary and at the clinic visits.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany

REFERENCES:
- [Result] Ziegler D, Hidvegi T, Gurieva I, Bongardt S, Freynhagen R, Sen D, Sommerville K; Lacosamide SP743 Study Group. Efficacy and safety of lacosamide in painful diabetic neuropathy. Diabetes Care. 2010 Apr;33(4):839-41. doi: 10.2337/dc09-1578. Epub 2010 Jan 12. PMID 20067958